CLINICAL TRIAL: NCT01586663
Title: Evaluation of Serial Night Time Position Splint on Range of Motion for Patients With Systemic Sclerosis
Brief Title: Serial Night Time Position Splint on Systemic Sclerosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Fernanda Pontes Cardoso, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP 1070/09
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Diffuse Systemic Sclerosis
Keywords: Diffuse Systemic Sclerosis; Hand; Range of motion; Splint
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): Splint group
  Interventions: Device: Serial night time position splint
- Control Group (Active Comparator): Drug treatment
  Interventions: Drug: Drug treatment

INTERVENTIONS:
Device: Serial night time position splint — This group will use a serial night time position splint, adjusted monthly, during three months.
  Arms: Experimental Group
Drug: Drug treatment — This patients will keep there drug treatment and will receive their splints on the end of the study.
  Arms: Control Group

SUMMARY:
This is a randomized controlled trial with blinded evaluator and follow-up of one year. Seventy six patients with diffuse systemic sclerosis, will be randomized into two groups.The patients can not change their medication during the study. Patients will be evaluated at baseline and at 3, 6, 9 and 12 months. The experimental group will use a serial night time position splint who will be adjusted monthly, while the control group will remain the drug treatment. The outcomes assessed will be: pain, hand range of motion, quality of life, functional capacity, upper limb function and dexterity. Our hypothesis is that the serial night time position splint will improve the hand range of motion in diffuse systemic sclerosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Diffuse Systemic scleroses diagnosed following the ACR criteria
* Older than 18 years old
* Sclerodactyly

Exclusion Criteria:

* Neurological, psychiatric diseases and other rheumatic disease (including overlapping)
* Previous use of splints or allergy to splint material
* Surgery schedule to the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Change in hand range of motion | Baseline and after 3, 6, 9 and 12 months
  Measured by goniometry

SECONDARY OUTCOMES:
Change in pain | Baseline, after 10, 20 and 40 weeks
  Measured by a visual analogue scale
Change in functional capacity | Baseline, after 10, 20 and 40 weeks
  Measured by HAQ questionnaire
Change in quality of life | Basline, after 10, 20 and 40 weeks
  Measured by SF-36 questionnaire
Change in upper limb function | Baseline, after 10, 20 and 40 weeks
  Measured by DASH questionnaire
Change in dexterity | Baseline, after 3, 6, 9 and 12 months
  Measured by SODA test

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Natour, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil